CLINICAL TRIAL: NCT00502138
Title: A Pilot Study to Assess the Pharmacokinetics, Pharmacodynamics and Safety/Tolerability of Pramlintide Acetate When Administered by Subcutaneous Infusion in a Basal-Bolus Manner as an Adjunct to Continuous Subcutaneous Insulin Infusion Therapy in Patients With Type 1 Diabetes
Brief Title: A Pilot Study of Continuous Subcutaneous Pramlintide Infusion Therapy in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Diabetes & Endocrine Consultants (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, David M. Huffman MD, Principal Investigator, University Diabetes & Endocrine Consultants
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pramlintide Infusion in IDDM
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: IDDM
Keywords: diabetes; insulin; pramlintide; IDDM
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — pramlintide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Interventional, continuous pramlintide infusion at 9 micrograms/hr plus 60 microgram meal bolus plus continuous insulin basal-bolus subcutaneous infusion
  Interventions: Drug: Continuous Pramlintide infusion

INTERVENTIONS:
Drug: Continuous Pramlintide infusion — pramlintide injection, 9 mcg/hr plus 60 mcg premeal boluses
  Other Names: pramlintide

SUMMARY:
This research project will investigate the effects of pramlintide (Symlin) given by continuous subcutaneous (under the skin) infusion throughout the day and night, along with meal doses similar to those injected during conventional pramlintide (Symlin) treatment, delivered using a second insulin pump, in subjects with inadequately controlled type I diabetes mellitus who are already using insulin pump therapy. Study participants will wear two pumps for a four month period, taking insulin in their usual manner and pramlintide (Symlin) in a similar basal/bolus fashion. Continuous glucose monitors will be worn on three occasions during the study to assess blood glucose responses to continuous pramlintide (Symlin) treatment.

DETAILED DESCRIPTION:
DESCRIPTION OF STUDY:

To participate in the study, you must have Type I diabetes mellitus and be taking insulin using an insulin pump, and have a hemoglobin A1c level between 7.0% and 10.0%. You will not be permitted to participate in the study if you have taken pramlintide (Symlin) during the previous three months. The study will consist of seven visits to the Study Center over a four-month period. Subjects will undergo meal tolerance testing at beginning and end of study period. Continuous blood glucose monitoring will be performed on three occasions during the study.

Pramlintide will be begun at a single basal rate of 1.5 units/hr. Bolus therapy will be begun thereafter per standard manufacturer protocol. Subjects will be monitored for three months on basal-bolus pramlintide therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes of at least one year duration;
2. Treated with CSII therapy for at least 6 months;
3. Age 18 to 70 years, inclusive;
4. A1C >7.0 and ≤10% as screening;
5. BMI ≤35 kg/m2;
6. Stable insulin dose (±10%) for at least 3 months prior to screening;
7. If female, has a negative urine pregnancy test at screening;
8. If female and of childbearing potential, practicing and willing to continue to using appropriate contraception to ensure that pregnancy does not occur during the study;
9. Able to understand and sign the required study documents and comply with the protocol requirements

Exclusion Criteria:

1. Is poorly compliant with the currently prescribed insulin regimen, as determined by the investigator;
2. Has any significant medical condition, laboratory findings, or medical history that may affect successful completion of the study and/or personal well-being;
3. If female and if of childbearing potential, is pregnant, lactating, or planning to become pregnant;
4. Has experienced recurrent severe hypoglycemia requiring assistance during the past 6 months;
5. Has a history of hypoglycemia unawareness;
6. Has a confirmed diagnosis of gastroparesis;
7. Requires the use of drugs that stimulate gastrointestinal motility;
8. Is receiving medications known to interfere with glycemic control (i.e. glucocorticoids);
9. Has been treated with any oral antidiabetic agent or exenatide within 3 months of screening visit;
10. Has been treated with pramlintide within 3 months of screening visit;
11. Has received an investigational drug within 3 month of screening visit;
12. Is currently participating in a clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Fasting and postprandial pramlintide pharmacokinetics | Four months

SECONDARY OUTCOMES:
Hemoglobin A1c, body weight, blood glucose variability, patient satisfaction | four months
Hemoglobin A1c | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David M Huffman, MD, Principal Investigator — University Diabetes & Endocrine Consultants
Locations (1):
- University Diabetes & Endocrine Consultants, Chattanooga, Tennessee, United States

REFERENCES:
- [Derived] Huffman DM, McLean GW, Seagrove MA. Continuous subcutaneous pramlintide infusion therapy in patients with type 1 diabetes: observations from a pilot study. Endocr Pract. 2009 Nov-Dec;15(7):689-95. doi: 10.4158/EP09044.ORR1. PMID 19546056